CLINICAL TRIAL: NCT02644811
Title: Miniscrews as Anchorage Device for Orthodontic Treatment - Randomized Controlled Trials on Anchorage Capacity, Cost Efficiency and Patient Acceptance
Brief Title: Miniscrews as Anchorage Device for Orthodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Gävleborg (Other)
Collaborators: Malmö University (Other); Department of Research and Development, County Council of Gavleborg and Uppsala University (Unknown); Swedish Dental Associations Scientific Funds (Unknown); Thuréus Foundation for the Promotion of Dental Science, Uppsala University, Sweden (Unknown)
Responsible Party: Principal Investigator, Niels Ganzer, DDS, Senior Consultant Orthodontist, Region Gävleborg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CFUG-479851
Record Dates: First submitted 2015-12-18; First posted 2016-01-01 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Orthodontic Anchorage Procedures; Orthodontic Space Closure
Keywords: Miniscrew; Temporary anchorage device (TAD); mini-implants; Miniscrew implant (MSI)
MeSH Terms: interventions — Anesthesia; Anesthesia, Local; Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A - Miniscrews (Experimental): Topical anesthesia (buccal and palatal) followed by local anesthesia (buccal and palatal). Extraction of the maxillary first premolars.
  Fixed appliance in the maxilla or maxilla and mandible.
  Anchorage reinforcement with miniscrews (Spider Screw K1 short neck). Miniscrews are placed buccally between the maxillary second premolar and the first molar after topical anesthesia (buccal) and injection (buccal). Miniscrews are placed when space closure starts. Space closure is performed as en masse retraction. Miniscrew are immediately loaded with 150g Nickel Titanium coil springs.
  Interventions: Drug: Topical anesthesia (buccal and palatal); Drug: Local anesthesia (buccal and palatal); Procedure: Extraction of the maxillary first premolars; Drug: Topical anesthesia (buccal); Drug: Local anesthesia (buccal); Device: Spider Screw K1 short neck
- Group B - Molarblock (Active Comparator): Topical anesthesia (buccal and palatal) followed by local anesthesia (buccal and palatal. Extraction of the maxillary first premolars.
  Fixed appliance in the maxilla or maxilla and mandible.
  Anchorage reinforcement with molarblocks - a Stainless steel ligature connecting the maxillary second premolar with the maxillary first and second molar. Molarblocks are installed from the beginning of leveling and alignment. Space closure is performed as en masse retraction with type one active tie-backs.
  Interventions: Drug: Topical anesthesia (buccal and palatal); Drug: Local anesthesia (buccal and palatal); Procedure: Extraction of the maxillary first premolars; Device: Molarblock

INTERVENTIONS:
Drug: Topical anesthesia (buccal and palatal) — Saliva is removed with a sterile swab followed by application of 5% Lidocaine gel (APL, Sweden) on the gingiva.
  Other Names: Anesthesic Jelly (buccal and palatal)
Drug: Local anesthesia (buccal and palatal) — Injection of 1,5 ml Xylocaine Dental Adrenaline (Lidocaine hydrochloride 20 mg/ml, adrenaline 12.5 µg/ml, Dentsply Pharmaceutical, Weybridge, Surrey, UK).
  Other Names: Injection (buccal and palatal)
Procedure: Extraction of the maxillary first premolars — Careful extraction of the maxillary first premolars after mobilization.
Drug: Topical anesthesia (buccal) — Saliva is removed with a sterile swab followed by application of 5% Lidocaine gel (APL, Sweden) on the gingiva.
  Other Names: Anesthesic Jelly (buccal)
  Arms: Group A - Miniscrews
Drug: Local anesthesia (buccal) — Injection of 0.3 ml Xylocaine Dental Adrenaline (Lidocaine hydrochloride 20 mg/ml, adrenaline 12.5 µg/ml, Dentsply Pharmaceutical, Weybridge, Surrey, UK).
  Other Names: Injection (buccal)
  Arms: Group A - Miniscrews
Device: Molarblock — Molarblock is a Stainless steel ligature connecting the maxillary second premolar with the maxillary first and second molar.
  Arms: Group B - Molarblock
Device: Spider Screw K1 short neck — The Spider Screw K1 (Health Development Company, Sarcedo, Italy) is a self-drilling and self-tapping screw. Short neck screws (SCR-1508 and SCR-1510) with a diameter of 1.5 mm and length 8 or 10 mm are used.
  Other Names: Temporary anchorage device; TAD; Orthodontic mini-implant
  Arms: Group A - Miniscrews

SUMMARY:
The purpose of this trial is to study and compare two different anchorage techniques. Adolescent patients in need for orthodontic treatment are randomized into Group A and B. Both groups are treated with extractions of the maxillary first premolars and fixed appliance. Anchorage is reinforced by miniscrews in Group A and by molarblock in Group B.

The hypotheses are:

* that placement of miniscrews does not cause more pain or discomfort than premolar extractions
* that molarblock provides increase of anchorage
* that miniscrews have a better anchorage capacity than molarblock
* that miniscrews are more cost-efficient than conventional anchorage techniques

DETAILED DESCRIPTION:
Participants are recruited from the orthodontic specialist clinic in Gävle, Sweden. After informed consent participants are randomized into Group A and B. The treatment starts with extractions of the maxillary first premolars. Extractions are performed by the participants´ general practitioner. Orthodontic treatment starts after the tooth extractions.

All participants get treatment with fixed appliance according to the straight wire concept (3M Victory brackets, .022 slot size, McLaughlin-Bennet-Trevesi prescription). The recommended wire sequence is: .016 Heat Activated Nickel Titanium, .019x.025 Heat Activated Nickel Titanium, .019x.025 Stainless Steel. Treatment time is about two years.

The following measurements are taken at:

T0 (Before treatment start): Study models, baseline questionnaire,

T1 (after tooth extractions, before the orthodontic treatment): Study models, cephalographic x-ray, questionnaire at the evening after tooth extractions, questionnaire one week after tooth extractions.

T2 (After miniscrew placement (Group A), Before space closure): Study models, cephalographic x-ray, questionnaire at the evening after miniscrew placement, questionnaire one week after miniscrew placement.

T3 (After space closure and miniscrew removal): Study models, cephalographic x-ray, questionnaire after screw removal

ELIGIBILITY:
Inclusion Criteria:

* Adolescents in need of orthodontic treatment with fixed appliance including extractions of the maxillary first premolars
* Need for Anchorage reinforcement
* Permanent dentition including the maxillary second molars in occlusion (DS4M2 according to Björk)
* Regular dental care in Sweden since the age of three.

Exclusion Criteria:

* Experience of previous orthodontic treatment
* Need for orthognathic surgery
* Need for maximum anchorage.

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Change in Tooth Position of the Maxillary Molars During Space Closure | Through Space Closure (T2-T3), an average of 9 months
  Tooth movement is assessed in millimeters using superimposition of study models and lateral cephalograms.

SECONDARY OUTCOMES:
Experience of Pain and Discomfort | Baseline, the evening after tooth extractions, one week after tooth extractions, the evening after miniscrew placement, one week after miniscrew placement
  Experiences of pain and discomfort are examined with validated self-report questionnaires.
Change in Tooth Position of the Maxillary Molars During Levelling and Alignment | Through Levelling and Alignment (T1-T2), an average of 9 months
  Tooth movement is assessed in millimeters using superimposition of study models and lateral cephalograms.
Societal Costs | Through Study Completion, an average of 2 years
  Societal costs are the sum of direct and indirect treatment costs. Direct costs are treatment time in the clinic and used material. Indirect costs are travel costs and costs for parents following the participant to the clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bondemark, Professor, Study Chair — Malmö University
Locations (1):
- Specialisttandvården Ortodonti, Gävle, Gävleborg County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feldmann I, List T, John MT, Bondemark L. Reliability of a questionnaire assessing experiences of adolescents in orthodontic treatment. Angle Orthod. 2007 Mar;77(2):311-7. doi: 10.2319/0003-3219(2007)077[0311:ROAQAE]2.0.CO;2. PMID 17319767
- [Background] Upadhyay M, Yadav S, Nanda R. Biomechanics of incisor retraction with mini-implant anchorage. J Orthod. 2014 Sep;41 Suppl 1:S15-23. doi: 10.1179/1465313314Y.0000000114. PMID 25138361
- [Background] Upadhyay M, Yadav S, Patil S. Mini-implant anchorage for en-masse retraction of maxillary anterior teeth: a clinical cephalometric study. Am J Orthod Dentofacial Orthop. 2008 Dec;134(6):803-10. doi: 10.1016/j.ajodo.2006.10.025. PMID 19061808
- [Background] Lehnen S, McDonald F, Bourauel C, Baxmann M. Patient expectations, acceptance and preferences in treatment with orthodontic mini-implants. A randomly controlled study. Part I: insertion techniques. J Orofac Orthop. 2011 Mar;72(2):93-102. doi: 10.1007/s00056-011-0013-8. English, German. PMID 21503849
- [Background] Feldmann I, List T, Feldmann H, Bondemark L. Pain intensity and discomfort following surgical placement of orthodontic anchoring units and premolar extraction: a randomized controlled trial. Angle Orthod. 2007 Jul;77(4):578-85. doi: 10.2319/062506-257.1. PMID 17605489
- [Background] Feldmann I, List T, Bondemark L. Orthodontic anchoring techniques and its influence on pain, discomfort, and jaw function--a randomized controlled trial. Eur J Orthod. 2012 Feb;34(1):102-8. doi: 10.1093/ejo/cjq171. Epub 2011 Feb 7. PMID 21300723
- [Background] Melsen B, Costa A. Immediate loading of implants used for orthodontic anchorage. Clin Orthod Res. 2000 Feb;3(1):23-8. doi: 10.1034/j.1600-0544.2000.030105.x. PMID 11168281
- [Background] Lai EH, Yao CC, Chang JZ, Chen I, Chen YJ. Three-dimensional dental model analysis of treatment outcomes for protrusive maxillary dentition: comparison of headgear, miniscrew, and miniplate skeletal anchorage. Am J Orthod Dentofacial Orthop. 2008 Nov;134(5):636-45. doi: 10.1016/j.ajodo.2007.05.017. PMID 18984395
- [Background] Papadopoulos MA, Tarawneh F. The use of miniscrew implants for temporary skeletal anchorage in orthodontics: a comprehensive review. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 May;103(5):e6-15. doi: 10.1016/j.tripleo.2006.11.022. Epub 2007 Feb 21. PMID 17317235
- [Derived] Ganzer N, Feldmann I, Petren S, Bondemark L. A cost-effectiveness analysis of anchorage reinforcement with miniscrews and molar blocks in adolescents: a randomized controlled trial. Eur J Orthod. 2019 Mar 29;41(2):180-187. doi: 10.1093/ejo/cjy041. PMID 30668660
- [Derived] Ganzer N, Feldmann I, Bondemark L. Anchorage reinforcement with miniscrews and molar blocks in adolescents: A randomized controlled trial. Am J Orthod Dentofacial Orthop. 2018 Dec;154(6):758-767. doi: 10.1016/j.ajodo.2018.07.011. PMID 30477773